CLINICAL TRIAL: NCT06043401
Title: Tracking Brain Biomarkers and Renormalization Associated With Antidepressant Transcranial Magnetic Stimulation Therapy
Acronym: INSCAPE
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Andrew Manett, Assistant Professor, Medical University of South Carolina
Other Study IDs: Pro00127417
Record Dates: First submitted 2023-08-16; First posted 2023-09-21 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Neuroimaging; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy volunteers: Age and sex-matched healthy individuals will also be recruited as a control group. They will be scanned three times (baseline, 3-week, and 6-week time points).
  Interventions: Other: Neuroimaging with Magnetic Resonance Imaging (MRI)
- volunteers with Major Depressive Disorder: 20 patients with MDD receiving standard-of-care depression treatment (TMS) at twill be recruited to participate in this observational neuroimaging study. They will be scanned three times (baseline, 3-week, and 6-week time points).
  Interventions: Other: Neuroimaging with Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Other: Neuroimaging with Magnetic Resonance Imaging (MRI) — MRI will be used to observe brain states over time.

SUMMARY:
This study will attempt to use magnetic resonance imaging (MRI) to take a picture of the brain to learn about changes that occur in the brain during Transcranial Magnetic Stimulation (TMS) in people receiving this treatment for depression.

DETAILED DESCRIPTION:
The purpose of this study is to take a picture of the participants brain using magnetic resonance imaging (MRI) and then use an investigational way of imaging the brain, called Individualized Network-based Single-frame Coactivation Pattern Estimation ("INSCAPE") to capture the participants brain activity. This method uses a computer program to understand which parts of the participants brain communicate with each other and creates a map of the brain areas that are connected.

The participants may take part in this study either because they are planning to receive Transcranial Magnetic Stimulation ("TMS") for Major Depressive Disorder ("MDD"), or because they are healthy volunteers. If the participants agree to take part in the study, they will attend three experimental visits in which they will undergo MRI scans. The interval between each experimental visits is about 3 weeks. The study itself does not provide TMS treatments, as it is only to attempt to observe the effects of TMS on the brain.

During each experimental visit, the investigators will conduct a brain scan for about 30 minutes in total. During the MRI scan, the participants will need to stay still, relax, and keep eyes open in the scanner. The purpose of this study is to explore whether this investigational brains can protocol, referred to as INSCAPE, can detect brain changes over the course of depression treatment while patients are receiving TMS. This method uses a computer program to understand which parts of the participants brain communicate with each other and creates a map of the brain areas that are connected.

ELIGIBILITY:
MDD volunteers:

Inclusion Criteria

* Age 18-65
* Have the capacity and ability to provide one's own consent in English and sign the informed consent document.
* DSM-IV diagnosis of MDD

Exclusion Criteria

* Unable to speak English.
* Contraindicated for MRI.
* Any current or recent untreated medical, neurological, or psychiatric conditions other than MDD that would preclude candidacy for TMS.
* Metal implant devices in the head, heart, or neck.
* History of brain surgery.
* History of cortisol medication use or electroconvulsive therapy.
* History of myocardial infarction or arrhythmia, bradycardia.
* Personal history of recent head injury, concussion, or self-report of moderate to severe traumatic brain injury.
* Individuals suffering from frequent/severe headaches.
* Moderate to severe alcohol or substance use disorder.
* Pregnancy

Healthy Volunteers Inclusion Criteria

* Age 18-65
* Have the capacity and ability to provide one's own consent in English and sign the informed consent document.

Exclusion Criteria

* Unable to speak English.
* Contraindicated for MRI.
* Any current or recent untreated medical, neurological, or psychiatric conditions
* Metal implant devices in the head, heart, or neck.
* History of brain surgery.
* History of cortisol medication use or electroconvulsive therapy.
* Comorbidity with other psychiatric/neurological illnesses or personality disorders
* History of myocardial infarction or arrhythmia, bradycardia.
* Personal history of recent head injury, concussion, or self-report of moderate to severe traumatic brain injury.
* Individuals suffering from frequent/severe headaches.
* Moderate to severe alcohol or substance use disorder.
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twenty patients with MDD receiving standard-of-care TMS treatment at the MUSC Brain Stimulation Service will be recruited to participate in this prospective neuroimaging study. No preference will be given based on race, gender, or ethnicity. Pregnant females and children under the age of 18 will be excluded for safety reasons. No vulnerable populations or special classes of subjects will be considered for participation.
  Twenty healthy controls will be enrolled as a comparison group.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Monitoring brain state renormalization with MRI | Baseline, 3-weeks, and 6-weeks, assessed up to 6 weeks.
  We will collect 3 MRI over the course of 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Manett, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT06043401/Prot_000.pdf
  • Informed Consent Form (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/01/NCT06043401/ICF_001.pdf